CLINICAL TRIAL: NCT05653024
Title: A Double-blind Randomized Controlled Trial of Inhaled Salbutamol vs Placebo for the Treatment of Acute Abdominal Pain From Food-induced IgE-mediated Reactions
Brief Title: INhaled Salbutamol vs Placebo for the Treatment of Acute IgE-mediated Abdominal Pain From Allergic Food REactions
Acronym: INSPIRE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was stopped due to unforseen changes in clinical practice (new oral immunotherapy focus on infants and toddlers) which led to a decrease in eligible participants and failure to meet recruitement targets.
Sponsor: Philippe Bégin (Other)
Responsible Party: Sponsor-Investigator, Philippe Bégin, Associate professor, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CITO-2022-01
Record Dates: First submitted 2022-11-22; First posted 2022-12-15 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: IgE-mediated Abdominal Pain
Keywords: food allergy; anaphylaxis
MeSH Terms: conditions — Food Hypersensitivity; Anaphylaxis | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled salbutamol (Experimental): 8 puffs of 100 mcg of inhaled salbutamol once
  Interventions: Drug: Salbutamol
- Placebo (Placebo Comparator): 8 puffs of inhaled placebo once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salbutamol — 8 puffs of 100 mcg inhaled salbutamol administered with spacer
  Other Names: Albuterol
  Arms: Inhaled salbutamol
Drug: Placebo — 8 puffs of placebo inhaler administered with spacer
  Arms: Placebo

SUMMARY:
The goal of this study is to assess the efficacy of inhaled salbutamol to treat abdominal pain during food allergic reactions.

Patients experiencing abominal pain as a result of a food allergic reaction during a food challenge in the allergy clinic will be invited to participate to the study.

They will receive either 8 puffs of salbutamol (asthma inhaler) or 8 puffs of a placebo inhaler.

The abdominal pain will then be followed using a numeric scale to see if patients receiving the medication experienced a faster improvement compared to those receiving the placebo.

DETAILED DESCRIPTION:
This trial aims to compare the efficacy of inhaled salbutamol compared to placebo to decrease the duration of abdominal pain in children and adults with IgE-mediated food allergic reactions.

The population will be children and adults aged 6 to 55 presenting with moderate to severe IgE-mediated abdominal pain in the context of an oral food challenge or an oral immunotherapy dose increase at the allergy clinic.

Eligible participants will be randomized to receive an immediate treatement with either inhaled salbutamol 800 mcg or inhaled placebo, dispensed with a spacer, at a ratio of 1:1.

Participants will be asked to rate the evolution of their abdominal pain by the minute on the NRS-11 scale until it resolves completely or that they have been discharged.

Patients still presenting moderate to severe abdominal pain 30 minutes after the administration of the investigational product will receive an open-label treatment with 800 mcg of inhaled salbutamol.

The primary outcome is the time from treatment to a decrease of the abdominal pain down to a mild intensity (defined as a pain for which the patient would not normally seek treatment).

Participants will be contacted by phone after three days to document any adverse event.

The primary endpoint will be analysed using a log-rank test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 6 to 55 years old.
* Undergoing an oral food challenge or an oral immunotherapy up-dosing visit for the diagnosis or treatment of an IgE-mediated food allergy.
* Previous confirmation of the food allergy by either skin prick tests (SPT) or serum specific IgE;
* Able to express the intensity of their pain using the NRS-11;
* Willing to comply with all study requirements.

Exclusion Criteria:

* Previous adverse reactions to salbutamol;
* Known hypersensitivity to salbutamol or placebo or any of their components;
* Any condition that could be considered a relative contra-indication to the use of salbutamol according to the investigator (e.g. patient with a history of hyperglycemia, arrhythmia or hypokalemia);
* Patients receiving beta-blockers or a daily / long-acting beta agonists;
* Patients needing to pass an anti-doping test for high-level sport in the following 24h.

Ages: 6 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Time to resolution of moderate-to-severe abdominal pain | From time of administation of investigational product, until the pain decreases to a point where the patient would not normally seek treatment, assessed up to 30 minutes
  Time from treatment to an abdominal pain of less than moderate intensity, defined as a pain for which the patient would not normally seek treatment

SECONDARY OUTCOMES:
Time to complete resolution of the abdominal pain | From time of administation of investigational product, until the pain is completely resolved, assessed up to 30 minutes
  Time from treatment to the complete resolution of the abdominal pain.
Time to any improvement in the abdominal pain | From time of administation of investigational product, until any decrease in the NRS-11, assessed up to 30 minutes
  Time from treatment to any decrease in the 11-point numeric pain rating scale (NRS-11)
Epinephrine use | From randomization to three days after randomization
  Overall rate of epinephrine administration following randomization
Adverse events | From randomization to three days after randomization
  Overall rate of adverse events following randomization

OTHER OUTCOMES:
Time to resolution of moderate-to-severe abdominal pain after open-label rescue | From time of administation of open-label rescue treatment, until the pain decreases to a point where the patient would not normally seek treatment, assessed up to patient discharge
  Time from open-label rescue treatment to an abdominal pain of less than moderate intensity, defined as a pain for which the patient would not normally seek treatment
Time to resolution of abdominal pain after open-label rescue | From time of administation of open-label rescue treatment, until complete resolution of the abdominal pain, assessed up to patient discharge
  Time from open-label rescue treatment to complete resolution of abdominal pain
Time to any improvement in abdominal pain after open-label rescue | From time of administation of open-label rescue treatment, until any decrease in the NRS-11, assessed up to patient discharge
  Time from open-label rescue treatment to any decrease in the NRS-11

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bégin, MD PhD, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Available upon request to corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: Protocol and SAP will be provided as supplementary material at time of study publication.
Access Criteria: As per journal policy